CLINICAL TRIAL: NCT01625390
Title: A Phase 2/3, Multicenter, Open-label Clinical Study to Assess the Safety and Efficacy of BAY86-6150 in Subjects With Hemophilia A or B With Inhibitors, Composed of 2 Parts (A & B). Part A: Sequential Cohorts of Four Dose Levels of the Modified rFVIIa BAY86-6150 Assessed in a Non-controlled Dose Response Design in Acutely Bleeding Subjects and for PK/ PD in an Intra-individual Crossover Design Compared With One Fixed Dose of Eptacog Alfa in Non-bleeding Subjects. Part B: Confirmatory Study to Further Investigate the Efficacy and Safety of BAY86-6150
Brief Title: A Phase 2/ 3 Trial to Evaluate the Efficacy and Safety of BAY86-6150
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15534; 2011-000323-33 (EudraCT Number); U1111-1133-2156 (Other: WHO - Universal Trial Number (UTN))
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Hemophilia A, Hemophilia B
Keywords: hemophilia, haemophilia, inhibitor, FVIIa, Factor VII activated, bypassing
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — Factor VII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: BAY86-6150
- Arm 2 (Active Comparator)
  Interventions: Drug: eptacog alfa [activated]
- Arm 3 (Experimental)
  Interventions: Drug: BAY86-6150

INTERVENTIONS:
Drug: BAY86-6150 — Four dose levels (6.5 µg/kg, 20 µg/kg, 50 µg/kg and 90 µg/kg) of BAY86-6150 will be studied.
  Arms: Arm 1
Drug: eptacog alfa [activated] — comparative PK/PD (pharmacokinetics/pharmacodynamics) evaluation
  Arms: Arm 2
Drug: BAY86-6150 — Confirmation of recommended dose of BAY86-6150 to be evaluated further as determined in Part A.
  Arms: Arm 3

SUMMARY:
Haemophilia is a disorder, usually genetic, affecting mostly male individuals, in which one of the proteins needed to form blood clots (FVIII) is missing or not present in sufficient levels. In a person with haemophilia, the clotting process is much slower and the person experiences bleeding episodes that can result in serious problems and potential disability.

The current haemophilia standard of care is to maintain FVIII activity level above 1%. Sometimes, patients can develop antibodies (so called "inhibitors") against FVIII and it is no longer effective at controlling bleeds. Bleeds in these patients are currently treated using other proteins involved in the clotting process.

The purpose of this study is to investigate how effectively BAY86-6150 may stop acute bleeds in "inhibitor" patients. This study consists of two parts, A and B. The purpose of part A is to find the most effective yet tolerable out of four doses of BAY86-6150 with regard to efficacy and safety (dose-finding part). Part A is expected to last 9 - 29 months. The purpose of part B is to confirm efficacy and safety of the dose found in part A in all participating patients (confirmatory part). Part B is expected to last 12-32 months.

Approximately 60 male subjects 12 to 62 years-of-age with moderate or severe haemophilia A or B, with inhibitors to FVIII or FIX, who have had 4 or more bleeding episodes in the last 6 months, will participate in this study.

Patient's bleeds will be treated with BAY86-6150 and with a rescue medication if no response is made to BAY86-6150. Patients will attend the treatment centre at regular intervals and be required to keep an electronic diary.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* 12 to 62 years-of-age
* History of moderate or severe congenital hemophilia A or B with inhibitors to FVIII or FIX
* 4 or more bleeding episodes in the last 6 months before enrollment.

Exclusion Criteria:

* Clinically relevant coagulation disorder other than congenital hemophilia A or B with inhibitors
* History of coronary and/or peripheral atherosclerotic disease
* Disseminated intravascular coagulopathy, or stage 2 hypertension
* Angina pectoris
* Myocardial infarction
* Transient ischemic attack
* Stroke
* Congestive heart failure
* Thromboembolic event

Ages: 12 Years to 62 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Successful treatments of bleeding episodes. | 10 hours after each bleed
  A bleed was defined as successfully treated, if no administration of rescue medication was required.
Proportion of successful treatments of bleeding episodes on subject level. | 10 hours after each bleed
  Proportion of successful treatments of bleeding episodes was calculated as number of bleeding episodes treated successfully - without rescue medication - divided by the total number of bleeding episodes on a dose level.

SECONDARY OUTCOMES:
Time to stop the bleed | 10 hours after each bleed
Number of injections needed to stop the bleeding episode. | 10 hours after each bleed
Effectiveness of treatment as rated by the subject's assessment (very effective, effective, partially effective, not effective). | 10 hours after each bleed
Participant's reported outcome as assessed by Euro QoL (EQ-5D). | 14 days after last exposure to BAY86-6150
Participant's reported outcome as assessed by Brief Pain Inventory. | 7 days after last exposure to BAY86-6150
Participant's reported outcome as assessed by Work Productivity and Activity Impairment Questionaire. | 14 days after last exposure to BAY86-6150

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (58):
- United States (2):
  - Sacramento, California
  - Chattanooga, Tennessee
- Melbourne, Victoria, Australia
- Brazil (2):
  - Rio de Janeiro, Rio de Janeiro
  - São Paulo, São Paulo
- Sofia, Bulgaria
- Santiago, Chile
- China (3):
  - Guangzhou, Guangdong
  - Beijing
  - Tianjin
- Colombia (2):
  - Barranquilla, Atlántico
  - Bogotá
- Aarhus N, Denmark
- France (2):
  - Lyon
  - Tours
- Germany (2):
  - Villingen-Schwenningen, Baden-Wurttemberg
  - Mainz, Rhineland-Palatinate
- Hungary (2):
  - Budapest
  - Debrecen
- India (4):
  - Hyderabad, Andhra Pradesh
  - Ludhiana, Punjab
  - Bangalore
  - Pune
- Tel Litwinsky, Israel
- Italy (2):
  - Florence
  - Milan
- Japan (3):
  - Kashihara, Nara
  - Shinjuku-ku, Tokyo
  - Suginami, Tokyo
- Mexico (4):
  - Guadalajara, Jalisco
  - Oaxaca City, Oaxaca
  - San Luis Potosí City, San Luis Potosí
  - México D. F.
- Utrecht, Netherlands
- Christchurch, New Zealand
- Warsaw, Poland
- Romania (2):
  - Timișoara, Timiș County
  - Bucharest
- Russia (4):
  - Khabarovsk
  - Saint Petersburg
  - Samara
  - Yekaterinburg
- Singapore, Singapore
- South Africa (3):
  - Bloemfontein, Freestate
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
- Seoul, South Korea
- Gothenburg, Sweden
- Taiwan (3):
  - Taipei, Taipei
  - Changhua
  - Taipei
- Turkey (Türkiye) (2):
  - Istanbul
  - Izmir
- Ukraine (3):
  - Donetsk
  - Lviv
  - Odesa
- United Kingdom (2):
  - London
  - Truro